CLINICAL TRIAL: NCT02370329
Title: Phase II Study of P1101 in Early Myelofibrosis
Brief Title: P1101 in Treating Patients With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug became commercially available
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC138F; NCI-2015-00183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC138F (Other: Mayo Clinic in Arizona); 14-001548 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2024-09

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PEG-proline-interferon alpha-2b) (Experimental): Patients receive PEG-proline-interferon alpha-2b SC on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Ropeginterferon Alfa-2B

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Ropeginterferon Alfa-2B — Given SC
  Other Names: AOP2014; Besremi; P-1101; P1101; PEG-P-IFN-Alfa-2b; PEG-P-IFN-Alpha-2b; PEG-Proline-Interferon Alfa-2b

SUMMARY:
This pilot phase II trial studies P1101 (polyethyleneglycol [PEG]-proline-interferon alpha-2b) in treating patients with myelofibrosis. PEG-proline-interferon alpha-2b is a substance that can improve the body's natural response and may slow the growth of myelofibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate for clinical response (complete remission [CR], partial remission [PR], or clinical improvement [CI]) as defined by International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria in a cohort of intermediate-2/high risk myelofibrosis (MF) patients. Response in a second cohort of early stage MF patients will also be described.

SECONDARY OBJECTIVES:

I. To evaluate the adverse event profile of P1101 in patients with myelofibrosis by cohort (early vs intermediate-2/high risk).

II. To evaluate the tolerability of P1101 in patients with myelofibrosis by cohort (early vs intermediate-2/high risk).

EXPLORATORY AND CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate quality of life (QOL) and patient-reported symptoms using the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) with P1101 for patients with myelofibrosis by cohort (early vs intermediate-2/high risk).

II. To evaluate the impact of P1101 on bone marrow and histological features of myelofibrosis including cytogenetics, blast percentage, fibrosis, and JAK2-V617F allele burden by cohort (early vs intermediate-2/high risk).

OUTLINE:

Patients receive PEG-proline-interferon alpha-2b subcutaneously (SC) on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Evaluable myelofibrosis by IWG-MRT criteria including one or more of the following:

  * Spleen >= 5 cm below the left costal margin
  * MPN-SAF total symptom score (TSS) > 10 at baseline
  * Hemoglobin < 10 g/dL
* Confirmed diagnosis of myelofibrosis (primary myelofibrosis or myelofibrosis secondary to essential thrombocythemia or polycythemia vera) by World Health Organization (WHO) diagnostic criteria (3 major and 2 minor criteria: major criteria: megakaryocyte proliferation and atypia with either reticulin and/or collagen fibrosis, not meeting criteria for chronic myelogenous leukemia [CML], polycythemia vera [PV], myelodysplastic syndrome [MDS], or other myeloid neoplasm, JAK2V617F or other clonal marker or no evidence of reactive marrow fibrosis; minor criteria: leukoerythroblastosis, increased lactate dehydrogenase [LDH], anemia, palpable splenomegaly)
* For cohort 1: early stage MF (low or intermediate 1 stage as defined by Dynamic International Prognostic Scoring System [DIPSS]) without currently available treatment options
* For cohort 2: intermediate-2 or high risk MF patients as defined by DIPSS either not eligible for ruxolitinib or having failed under ruxolitinib
* No prior treatment for myelofibrosis (for cohort 1 only)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 2.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to return to enrolling institution for follow-up
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Patients who have had chemotherapy or radiation =< 2 weeks of registration
* For cohort 1 only: patients with evidence of intermediate 2 or high risk disease (according to DIPSS)
* For cohort 1 only: patients with a bone marrow biopsy with < 15% cellularity, evidence of collagen fibrosis, osteosclerosis, or blasts > 10% in peripheral blood or marrow (demonstrating advanced disease)
* Patients who have received a prior stem cell transplant
* Patients who have received radiation to the spleen within 3 months prior to registration
* Patients with intolerance to compounds similar to pegylated interferon alpha-2b
* Patients with evidence of >= grade 2 peripheral sensory neuropathy
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients or patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Uncontrolled simultaneous illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, history of depression, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* History of significant or major funduscopic findings including, but not limited to, retinal exudates, hemorrhage, detachment, neovascularization, papilledema, optic atrophy, micro-aneurysm or macular changes
* Other active malignancy at time of registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Palmer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (PEG-proline-interferon alpha-2b): Patients receive PEG-proline-interferon alpha-2b SC on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients will be started at a dose level of 100 micrograms (mcg) every other week, and then dose will be titrated up by 50mcg increments to a maximum dose of 300mcg every other week as tolerated.
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Ropeginterferon Alfa-2B: Given SC
Period: Overall Study
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
Started | 11
Completed | 0
Not Completed | 11
Not completed — Alternate treatment | 1
Not completed — Adverse Event | 1
Not completed — Disease progression | 3
Not completed — Physician Decision | 2
Not completed — Study closure | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 69 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Myelofibrosis Risk Stage [Count of Participants; unit: Participants] — Scored according to the Dynamic International Prognostic Scoring System (DIPSS) for primary myelofibrosis.> Each of the following factors are assigned 1 point:>
  * age older than 65>
  * leukocyte count higher than 25x10^9L>
  * circulating blasts>=1%>
  * constitutional symptoms> The following is assigned 2 points:>
  * hemoglobin lower than 10 g/dL>
  Risk group:>
  * low (0 points)>
  * intermediate-1 (1-2 points)>
  * intermediate-2 (3-4 points)>
  * high (5-6 points)
  Participants
    Low/Intermediate-1 risk stage | 4
    Intermediate-2/high risk stage | 7
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction>
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work>
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours>
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours>
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair>
  5. Dead
  Participants
    0 | 8
    1 | 2
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (Complete Remission, Partial Remission, or Clinical Improvement) as Determined by International Working Group Criteria
Description: Patients will be assessed for response according to the Revised International Working Group for Myeloproliferative Neoplasms Research and Treatment criteria.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
Number analyzed (Participants) | 11
Participants
  Clinical Improvement | 7
  Stable Disease | 3
  Progression | 1

2. Secondary Outcome: Progression-free Survival Time
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
Number analyzed (Participants) | 11
months | NA [31.9 to NA] — The median and upper limit of the confidence interval were not reached due to a low number of events.

3. Secondary Outcome: Number of Patients Experiencing a Grade 3+ Adverse Event, as Measured by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4)
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
Number analyzed (Participants) | 11
Participants | 10

4. Other Pre Specified Outcome: Changes in Patient-reported Symptoms and QOL as Measured by MPN-SAF
Description: Patient-reported symptoms and QOL will be described at each time point using the mean, confidence interval, median, and range. Changes in individual symptoms, changes in a symptom scale composed of symptoms specific to MF patients, and changes in the MPN TSS will be investigated. Graphical procedures will include stream plots of individual patient scores and plots of average values over time. Correlational analyses will be done to determine the relationships among patients-reported symptoms and QOL, as well as with clinical outcomes and clinician-assessed symptoms.
Time Frame: Baseline to up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment (PEG-proline-interferon alpha-2b)
All-Cause Mortality (participants affected / at risk) | 3/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PEG-proline-interferon alpha-2b) (N=11)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PEG-proline-interferon alpha-2b) (N=11)
Anemia (Blood and lymphatic system disorders) | 9 (53)
Diarrhea (Gastrointestinal disorders) | 5 (39)
Nausea (Gastrointestinal disorders) | 3 (17)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders and administration site conditions) | 4 (21)
Sinusitis (Infections and infestations) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (36)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (57)
Platelet count decreased (Investigations) | 3 (40)
Weight loss (Investigations) | 3 (4)
White blood cell decreased (Investigations) | 8 (133)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (5)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (16)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02370329/Prot_SAP_000.pdf